CLINICAL TRIAL: NCT03910348
Title: Effects of Whole-Body Vibration and High Impact Exercises on the Bone Metabolism and Fall Risk in Postmenopausal Women
Brief Title: Effects of Whole-Body Vibration and High Impact Exercises in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ekin Ilke Sen, Medical doctor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IstanbulU-Ekin Sen
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Osteoporosis, Postmenopausal; Exercise Therapy
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whole body vibration exercise (Experimental): The WBV training consisted of a high frequency (30-40 Hz) vibration stimulus at a low setting (2-4mm peak to peak) on a Power Plate pro5 vibration platform (Performance Health Systems, LLC, Northbrook, IL, USA). Each patient received the vibrations under supervision using five different static positions: squat, deep squat, widestep squat, lunge, and hands-front lunge. The exercise programs for each experimental groups consisted of 20 to 60-minute sessions on three days per week for 24 weeks, and they were performed under the supervision.
  Interventions: Device: Whole-body vibration exercise
- High-impact exercise (Experimental): Depending on their individual calcium and vitamin D intakes, each patient advised to receive supplemental calcium and vitamin D to ensure a total daily intake of 1,500 mg of calcium and 880 IU of vitamin D.
  Interventions: Other: High-impact exercise
- Control (No Intervention): Depending on their individual calcium and vitamin D intakes, each patient received supplemental calcium and vitamin D to ensure a total daily intake of 1,500 mg of calcium and 880 IU of vitamin D. The demographic characteristics of the participants were obtained at the baseline assessment.

INTERVENTIONS:
Device: Whole-body vibration exercise — The WBV training consisted of a high frequency (30-40 Hz) vibration stimulus at a low setting on a Power Plate pro5 vibration platform (Performance Health Systems, LLC, Northbrook, IL, USA).
  Arms: Whole body vibration exercise
Other: High-impact exercise — In the high-impact exercise program, the patients were asked to jump using a jump-rope at the beginning of each session
  Arms: High-impact exercise

SUMMARY:
We investigated the effects of whole body vibration (WBV) and high-impact (HI) exercises in postmenopausal women with low bone mineral density. In summary, WBV exercises are effective in preventing bone loss and WBV and HI exercise programs are effective in decreasing fall risk, increasing health-related quality of life and improving depressive symptoms

DETAILED DESCRIPTION:
Purpose: The aim of this study was to determine the effects of six months of supervised whole-body vibration (WBV) and high-impact (HI) exercises on bone mineral density (BMD), serum bone turnover markers, fall risk, health-related quality of life (HRQoL) and depressive symptoms in postmenopausal women, additionally, to evaluate the advantage of each training program to another.

Methods: In a prospective, randomized controlled 6-month interventional trial 58 eligible postmenopausal women were assigned to WBV training group (n=19), HI training group (n=19), or control group (n=20). The patients in both training groups participated in a supervised training program, which consisted of the one-hour exercise session three times a week for six months. The WBV groups received vibration (30-35 Hz, 2-4 mm) in five different static positions. The HI group jumped rope (10-50 jumps/day). All patients received calcium (1000 mg) and vitamin D (880 IU) supplementation per day. In all participants, baseline and six-month BMD at the lumbar spine and femur were measured by Dual-energy X-ray Absorptiometry (DXA). Serum osteocalcin (OC) and C-terminal telopeptide of type I collagen (CTx) were measured at baseline, three- and six-month intervals. Fall risk was assessed by using the Timed Up and Go (TUG) test and fall index measured by static posturography at baseline, three- and six-month intervals. HRQoL and depressive symptoms were assessed using the Quality of Life Questionnaire of the European Foundation for Osteoporosis (QUALEFFO) and Beck Depression Inventory (BDI), respectively, at baseline and six-month of the study.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged 40-65 years old
* Bone mineral density T-scores between -2.0 and -3.0 at the L1-L4, L2-L4, femoral neck, trochanter and/or total hip regions
* Serum 25(OH)vitamin D level ≥ 30 ng/ml.

Exclusion Criteria:

* The use of any medications and/or disease that affect bone metabolism
* Neuromuscular performance, and/or balance; presence of cardiovascular, pulmonary, neuromuscular, and/or chronic diseases that affect exercise training
* Presence of an osteoporotic fracture
* Presence of a musculoskeletal disease, such as an acute lumbar herniated disc and/or spondylolisthesis
* Presence of gall or kidney stones, prostheses, intraocular lenses, and/or implants
* Body mass index ≥35 kg/m²
* Thrombosis history

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Bone Mineral Density at 6 months | baseline and 6 month
  The bone mineral density of the lumbar spine, femoral neck were measured with a dual energy x-ray absorptiometry

SECONDARY OUTCOMES:
Change from Baseline Bone Formation Marker at 3-months and 6-months | baseline, 3-month, 6-month
  The serum osteocalcin (OC) level
Change from Baseline Bone Resorption Marker- at 3-months and 6-months | baseline, 3-month, 6-month
  The serum C-terminal telopeptide of type I collagen (CTx) levels
Change from Baseline Fall risk at 3-months and 6-months | baseline, 3-month, 6-month
  A computerized static posturography device was used to measure the fall index
Change from Baseline Functional Balance at 3-months and 6-months | baseline, 3-month, 6-month
  Timed Up and Go (TUG) test
Change from Baseline Health-related Quality of Life at 6 months | baseline, 6-month
  Quality of Life Questionnaire of the European Foundation for Osteoporosis (QUALEFFO)
Change from Baseline Depressive Symptoms at 6 months | baseline, 3-month, 6-month
  Beck Depression Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Ekin I Sen, Principal Investigator — Istanbul University